CLINICAL TRIAL: NCT06356415
Title: Infraclavicular Brachial Plexus Block Using Bupivacaine Alone or in Combination With Dexmedetomidine and Dexamethasone for Hand and Forearm Surgeries, A Randomized, Controlled Trial
Brief Title: Infraclavicular Brachial Plexus Block With Bupivacaine Alone or With Both Dexmedetomidine and Dexamethasone
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Suez Canal University (Other)
Responsible Party: Principal Investigator, Abdelrhman Alshawadfy, Assistant Professor Suez Canal University Faculty of Medicine, Suez Canal University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Dex Dex in infraclavicular
Record Dates: First submitted 2024-04-04; First posted 2024-04-10 (Actual); Last update posted 2024-04-10 (Actual); Status verified 2024-04

CONDITIONS: Upper Extremity Injury
MeSH Terms: conditions — Arm Injuries | interventions — Bupivacaine

STUDY DESIGN:
Who Masked: Participant
Masking Description: The sealed-envelope technique will be used. An assistant who is not involved in patient care will make and combine bupivacaine, whether it contains adjuvants or not. Thus, all patients, operators, and outcome assessors remain blinded to the nature of the perineural adjuvant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bupivacaine (Active Comparator): Patients will undergo an ultrasound-guided infraclavicular brachial plexus block using bupivacaine alone.
  Interventions: Drug: Bupivacaine injection
- Bupivacaine+ Dexamethasone+ Dexmedetomidine (Active Comparator): Patients will undergo an ultrasound-guided infraclavicular brachial plexus block using bupivacaine combined with dexmedetomidine and dexamethasone.
  Interventions: Drug: Bupivacaine+ Dexamethasone+ Dexmedetomidine

INTERVENTIONS:
Drug: Bupivacaine injection — Group one will receive infraclavicular block using bupivacaine
  Arms: Bupivacaine
Drug: Bupivacaine+ Dexamethasone+ Dexmedetomidine — Group two will receive infraclavicular block using dexamethasone and dexmedetomidine added to the bupivacaine
  Arms: Bupivacaine+ Dexamethasone+ Dexmedetomidine

SUMMARY:
Upper-extremity regional anesthetic techniques, using brachial plexus blockade, have been shown to reduce adverse effects related to opioid administration, improve patient satisfaction, and provide significantly improved analgesia immediately following these surgeries. Many medications have been investigated to extend and enhance long-acting local anesthetics' (LA) analgesic effects. Currently, dexamethasone and dexmedetomidine have been studied, looking for an optimal long-lasting single-shot nerve block. In general, adjuvants have been used in peripheral nerve blocks to accelerate onset, decrease plasmatic absorption and secondary toxic effects, and prolong the block effects.

DETAILED DESCRIPTION:
Brachial plexus blockade-based upper-extremity regional anesthetic approaches have been demonstrated to lessen opioid administration side effects, increase patient satisfaction, and offer noticeably better analgesia right after these surgeries. A lot of drugs have been tested to prolong and improve the analgesic effect of long-acting local anesthetics (LA). Currently, dexamethasone and dexmedetomidine have been studied, looking for an optimal, long-lasting single-shot nerve block. Adjuvants have generally been employed in peripheral nerve blocks to lengthen the block effects, limit secondary toxic effects and plasmatic absorption, and speed the onset of the block. Objectives: To compare the effects of adding dexmedetomidine and dexamethasone to bupivacaine on the start of sensory blockade in an infraclavicular brachial plexus block. Patients and Methods: A prospective, randomized controlled trial will be conducted on patients who are undergoing hand or forearm surgeries. Patients who will be eligible for the study will be divided into 2 groups. The first group will receive dexmedetomidine and dexamethasone as adjuvants to bupivacaine, while the second group will receive bupivacaine alone. Expected Results: The success rate, onset time, duration of the block, and possible adverse events.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-65 years
* American Society of Anesthesiologists physical status I-II
* Body mass index between 18 and 35 kg/ m2
* scheduled for forearm and hand surgeries

Exclusion Criteria:

* Inability to consent to the study
* Coagulopathy
* Sepsis
* Decompensated chronic hepatic or renal illnesses
* Allergy to any of the used drugs
* Pre-existing musculocutaneous/median/radial/ ulnar neuropathy
* Prior surgery in the infraclavicular fossa

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-05-01 (Estimated); Primary Completion 2024-08-30 (Estimated); Study Completion 2024-09-30 (Estimated)

PRIMARY OUTCOMES:
Onset of sensory block | Immediately after the performance of the infraclavicular block
  Comparing the number of minutes required to achieve total upper limb sensory blockade following the application of an infraclavicular brachial plexus block that includes both dexmedetomidine and dexamethasone in addition to bupivacaine, as opposed to merely using bupivacaine on its own.